CLINICAL TRIAL: NCT02105376
Title: The Effects of Trigeminal Nerve Stimulation (TNS) for the Treatment of Major Depressive Disorder: a Phase II, Randomized, Sham Controlled Clinical Trial
Brief Title: TNS for Major Depressive Disorder: a Phase II Randomized Controlled Trial
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Santa Casa Medical School (Other)
Collaborators: Faculdade de Ciências Médicas da Santa Casa de São Paulo (Other)
Responsible Party: Principal Investigator, Pedro Shiozawa, Pedro Shiozawa, Coordinator, Laboratory of Clinical Neuromodulation, Principal Investigator, Faculdade de Ciências Médicas da Santa Casa de São Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TNS_depression
Record Dates: First submitted 2014-02-10; First posted 2014-04-07 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-05

CONDITIONS: Depressive Symptoms
Keywords: depression; cranial nerve stimulation; trigeminal stimulation
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Trigeminal Nerve Stimulation (TNS) (Experimental): TNS active group
  TNS will be applied by the external simulator EMS400. The stimulation will be conducted at a frequency of 120 Hz with pulse duration of 200 microseconds. The current intensity will be individually established and should be equivalent to a slight feeling of not painful paresthesia (approximately 0.5-2mA). The stimulus generates a pulse and asymmetric biphasic waveform. Electrodes (25cm2) will be placed on the forehead just above the supraorbital foramen bilaterally.
  Interventions: Device: Trigeminal Nerve Stimulation (TNS)
- Sham (Placebo Comparator): TNS sham
  The placebo intervention will consist of an initial stimulation until a mild paresthesia is achieved, and then turn off the machine after 60 seconds, after which period there is a tendency of reduction natural feeling secondary to skin sensitization paresthesia.

INTERVENTIONS:
Device: Trigeminal Nerve Stimulation (TNS) — Trigeminal Nerve Stimulation (TNS)
  Arms: Trigeminal Nerve Stimulation (TNS)

SUMMARY:
This is a phase II, randomized, sham controlled, clinical trial. This clinical trial has as primary objective to evaluate the effect of the Trigeminal Nerve Stimulation (TNS) on depressive symptoms measured by the Hamilton Depressive Rating Scale version 17 items (HDRS-17) in patients with moderate / severe depressive episode.

ELIGIBILITY:
Inclusion Criteria:

1. patients between 18 and 69 years
2. patients with a diagnosis of depression according to the SCID
3. score greater than or equal to 18 on the Hamilton Rating Scale 17-item version (equivalent to moderate or severe depressive episode)
4. agreement to participate in the study as recommended in the IC.

Exclusion Criteria:

1. patients with psychiatric indication for hospitalization
2. patients with psychiatric comorbidity
3. patients with a diagnosis of personality disorder
4. presence of severe neurological or medical diseases such as neoplasms in activity, neurodegenerative diseases and chronic diseases uncompensated.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2014-05; Primary Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Hamilton Depressive Rating Scale version 17 items (HDRS-17) | Change from baseline in depressive symptoms at 2 weeks
  This clinical trial has as primary objective to evaluate the effect of the Trigeminal Nerve Stimulation (TNS) on depressive symptoms measured by the Hamilton Depressive Rating Scale version 17 items (HDRS-17) in patients with moderate / severe depressive episode.

SECONDARY OUTCOMES:
Montreal Cognitive Assessment (MOCA) | Change from baseline in cognitive functioning at 2 weeks
  We also use the questionnaire Montreal Cognitive Assessment (MOCA) for assessment of cognitive function, considering the level of consciousness and global functioning in order to compare your score with estimates made by other instruments. It will also serve to assess possible cognitive damage and whether there are improvements in some specific cognitive functions with treatment

CONTACTS AND LOCATIONS:
Overall Officials: Quirino Cordeiro, MD, PhD, Study Director — Santa Casa Medical School; Pedro Shiozawa, MD, Principal Investigator — Santa Casa Medical School
Locations (1):
- Centro de Atencao Integrada à Saúde Mental, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Cook IA, Schrader LM, Degiorgio CM, Miller PR, Maremont ER, Leuchter AF. Trigeminal nerve stimulation in major depressive disorder: acute outcomes in an open pilot study. Epilepsy Behav. 2013 Aug;28(2):221-6. doi: 10.1016/j.yebeh.2013.05.008. Epub 2013 Jun 14. PMID 23773978
- [Background] DeGiorgio CM, Fanselow EE, Schrader LM, Cook IA. Trigeminal nerve stimulation: seminal animal and human studies for epilepsy and depression. Neurosurg Clin N Am. 2011 Oct;22(4):449-56, v. doi: 10.1016/j.nec.2011.07.001. PMID 21939843
- [Background] Schrader LM, Cook IA, Miller PR, Maremont ER, DeGiorgio CM. Trigeminal nerve stimulation in major depressive disorder: first proof of concept in an open pilot trial. Epilepsy Behav. 2011 Nov;22(3):475-8. doi: 10.1016/j.yebeh.2011.06.026. Epub 2011 Aug 4. PMID 21820361
- [Background] Shiozawa P, Cordeiro Q, Fregni F, Brunoni AR. Is sertraline plus transcranial direct current stimulation the future of effective depression treatment? J Comp Eff Res. 2013 May;2(3):213-5. doi: 10.2217/cer.13.28. No abstract available. PMID 24236617
- [Background] Riva-Posse P, Hermida AP, McDonald WM. The role of electroconvulsive and neuromodulation therapies in the treatment of geriatric depression. Psychiatr Clin North Am. 2013 Dec;36(4):607-30. doi: 10.1016/j.psc.2013.08.007. Epub 2013 Oct 6. PMID 24229660
- [Background] Vuilleumier P, Sander D, Baertschi B. Changing the brain, changing the society: clinical and ethical implications of neuromodulation techniques in neurology and psychiatry. Brain Topogr. 2014 Jan;27(1):1-3. doi: 10.1007/s10548-013-0325-7. Epub 2013 Oct 25. PMID 24158724